CLINICAL TRIAL: NCT02575248
Title: Induction of Ovulation by Clomiphene Citrate Following Laparoscopic Surgery for Endometriosis Stage 1 and Stage 11 With and Without Suppression by Dienogest
Brief Title: Induction of Ovulation by Clomiphene Citrate Following Laparoscopic Surgery for Endometriosis Stage 1 and Stage 2 With and Without Suppression by Dienogest
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alhassan Mohammad Khedr, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: fwa000017585
Record Dates: First submitted 2015-09-05; First posted 2015-10-14 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Infertility
Keywords: dienogest; infertility; endometriosis
MeSH Terms: conditions — Infertility; Endometriosis | interventions — dienogest; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): patients diagnosed laparoscopically with Endometriosis Stage 1 and Stage 2
  Interventions: Drug: Dienogest 2mg; Drug: Clomiphene citrate 5 mg
- group B (Active Comparator): patients diagnosed laparoscopically with Endometriosis Stage 1 and Stage 2
  Interventions: Drug: Clomiphene citrate 5 mg

INTERVENTIONS:
Drug: Dienogest 2mg — Dienogest 2mg is given daily for 3 months then followed by Clomiphene citrate 5 mg induction of ovulation for three months
  Arms: Group A
Drug: Clomiphene citrate 5 mg — Clomiphene citrate 5 mg for induction of ovulation for three months

SUMMARY:
This study aims at investigating the fertility outcome of endometriosis suppression with dienogest 2mg / day for 3 month followed by induction of ovulation for 3 month in endometriosis patients stage I and II.

DETAILED DESCRIPTION:
Study population: Sample size:

Group sample sizes of this study is 155 in group one and 155 in group two achieve 80% power to detect a difference between the group proportions of 0.10. The proportion in group one (the treatment group) is assumed to be 0.1000 under the null hypothesis and 0.2000 under the alternative hypothesis. The proportion in group two (the control group) is 0.1000. The test statistic used is .the one-sided Z test with un pooled variance. The significance level of the test was targeted at 0.05

Primary outcome:

Clinical pregnancy rate in endometriosis patients stage I and II undergoing endometriosis suppression with dienogest 2mg / day for 3 month followed by induction of ovulation for 3 month.

Secondary outcome:

Ovulation rate in endometriosis patients stage I and II undergoing endometriosis suppression with dienogest 2mg / day for 3 month followed by induction of ovulation for 3 month.

Inclusion criteria:

All women recruited in this study will have the have a definitive diagnosis of endometriosis grade I or grade II via laparoscopy just before randomization.

Method of Randomization:

A Computerized generated list from the internet https://www.sealedenvelope.com/sirnple-randomiser/vl/lists

Allocation concealment:

Closed envelope method by a nurse not participating in the study Intervention It is a prospective randomized controlled trial. Investigation done after recruitment and before randomization.

The patients will be randomized in to two groups:

Group A: patients receive dienogest 2 mg (visanne 2mg sanofi Aventis) daily for three months then followed by induction of ovulation with clomiphene citrate (clomid 5mg sanofi aventis for three months.

Group B: Patients will undergo induction of ovulation with clomiphene citrate (clomid 50mg sanofi aventis) for three months.

Protocol of induction of ovulation

1. Clomiphen citrate (clomid 50mg sanofi aventis) will be given on day two of the menstrual cycle at a dose of 50 mg twice daily for five days.
2. Folliculometry will be performed every other day starting from seventh day of the cycle till ovulation occurs using a 6 Mhz transvaginal probe till the follicles reach 18 - 20 mm.
3. A trigger of ovulation HCG 10000iu is given IM when the follicles reach 18- 22 mm. The couple will be advised to have intercourse after 36 hrs then daily for 7 days.
4. Prontogest 400 mg (progest 400 mg Sanofi Aventis) daily vaginal suppository as a luteal phase support.
5. Pregnancy will be diagnosed quantitative B HCG blood test after 2 days missed period.
6. Clinical pregnancy rate will be diagnosed by TVUS confirmed fetal echo with pulsation at 5-7 weeks gestation.

The sonographer confirming clinical pregnancy will be blinded to both groups. Statistical Analysis

Statistical Method:

Statistical analysis will be performed using Microsoft Excel version 2010 and statistical package for social sciences ( SPSS ) for windows version l S.O.

Continious data are to be presented as range, mean and standard deviation (if parametric); or range; median and inter quartile range (if non - parametric).

Dichotomous or categorical data are to be presented as number and percentage. Difference between independent is to be estimated using independent student's t-test (for parametric continuous variables), Manny whitney test U-test (for non -parametric continuous variables) and Chi-square and test (for categorical variables). Receiver operator characteristics curve is to be constructed to assess the predictability is to be expressed in terms of sensitivity , specificity , positive and negative predictive values. Significance level is at 0.05.

Ethical and legal aspects

Delegation of investigator responsibilities:

The investigator will ensure that all persons assisting with the trial are adequately informed about the protocol, any amendments to the protocol, the study treatments, and their trial-related duties and functions.

Patient information and informed consent:

Before being admitted to the clinical study, the patient must consent to participate after the nature, scope and possible consequences of the clinical study have been explained in a form understandable to her and a written consent will be obtained.

Confidentiality:

Only the patient initials will be recorded in the files, and if the patients name appears on any other document, it must be kept in a privacy by the investigators. The investigator will maintain a personal patient identification list (patient initials with the corresponding patient names) to enable records to be identified.

Protocol approval:

Before the beginning of the study and in accordance with the local regulation followed, the protocol and all the corresponding documents will be declared for Ethical and Research approval by the council of the obstetrics Department, Ain Shams University.

ELIGIBILITY:
Inclusion Criteria:

1. All women recruited in this study will have the have- a definitive diagnosis of endometriosis grade I or grade II via laparoscopy just before randomization.

Exclusion Criteria:

1. Male factor.
2. Other factors e.g. mullerian duct anomalies, hydrosalpinx.
3. Age > 35 years.
4. Day 3 FSH > 14 mlu/ml or antimullerian hormone <1 ng/1.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 2 months
  fetal life detected by ultrasound

SECONDARY OUTCOMES:
Ovulation rate | up to 21 days
  ovulation rate is recorded before triggering

CONTACTS AND LOCATIONS:
Overall Officials: laila fareed, lecturer, Study Director — 01222148471; mostafa fouad, professor, Study Director — 01226188993
Locations (1):
- AinShamsU, Abbasia, C, Egypt